CLINICAL TRIAL: NCT01598337
Title: The Effect Of Antiplatelets Therapy, Tirafiban, Prasugrel, And Aspirin On Saphenous Vein Coronary Artery Bypass Graft Patency
Brief Title: The Effect Of Antiplatelets Therapy On Saphenous Vein Coronary Artery Bypass Graft Patency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince Sultan Cardiac Center, Adult Cardiology Department. (Other)
Responsible Party: Principal Investigator, Abdulrahman Al-Moghairi, Principal Investigator, Prince Sultan Cardiac Center, Adult Cardiology Department.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSCC002CT
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Tirofiban; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aspirin alone (Active Comparator)
  Interventions: Drug: Aspirin; Drug: Tirofiban; Drug: Clopidogrel; Drug: Prasugrel
- Tirofoban (Experimental): Patient assigned to this arm will receive tirofiban infusion starting approximately six hours post bypass surgery once hemomstasis established and no evidence of bleeding
  Interventions: Drug: Tirofiban; Drug: Clopidogrel; Drug: Prasugrel
- Clopidogrel (Experimental): Patients receive oral clopidogrel 75 mg 6-8 hours before coronary bypass surgery and continue daily mentenance dose as per instruction by investigators
  Interventions: Drug: Tirofiban; Drug: Clopidogrel; Drug: Prasugrel
- Prasugrel (Experimental): Patients started on prasugrel 6 hours post surgery 10 mg then continue on daily 10mg as per instruction by investigators
  Interventions: Drug: Tirofiban; Drug: Clopidogrel; Drug: Prasugrel

INTERVENTIONS:
Drug: Aspirin — Patients continue their maintenance dose not inturrupted by surgery , 81 mg daily
  Arms: Aspirin alone
Drug: Tirofiban — Tirofiban infusion as specified by investigators to start after hemostasis been established
Drug: Clopidogrel — 75 mg orally started 6-8hours before surgery
Drug: Prasugrel — 10 mg daily as per instructions of investigators

SUMMARY:
This protocol is designed to evaluate the effect of antiplatelets (Tirafiban and Prasugrel) on the incidence of early and intermediate graft patency after CABG.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a commonly used revascularization strategy in patients with severe coronary artery disease. Saphenous vein grafts (SVGs) are the most frequently used conduits for this procedure. Unlike arterial grafts, SVGs are particularly susceptible to occlusive thrombosis during the first post-operative year, which exposes patients to increased risks of death, myocardial infarction, and repeat revascularization.

This study is designed to evaluate the effect of antiplatelets (Tirafiban and Prasugrel) on the incidence of early and intermediate graft patency after CABG. Patients will undergo planned cardiac Computed tomographic angiography (CTA) predischarge (at 1 week) and CTA/coronary angiography (CAG) at 6 months to 1 year follow-up. CTA at baseline (predischarge) and follow-up CTA/CAG at 6-12 months after CABG will be used to evaluate graft patency.

ELIGIBILITY:
Inclusion Criteria:

* All comer study where all patients undergoing coronary bypass surgery (CABG) will be randomized to one of the four treatment groups

Exclusion Criteria:

* Acute myocardial infarction (AMI) or cardiogenic shock
* Aortic dissection
* Mechanical valves.
* Contraindication to antiplatelets or aggrastat.
* Active bleeding or high risk of bleeding.
* History of hemorrhagic stroke any time.
* Recent history of embolic stroke or transient ischemic attack (TIA) less than 3 months.
* Active peptic ulcer disease (PUD).
* Liver derangement.
* Warfarin use.
* Heparin-induced thrombocytopenia (HIT) syndrome.
* Thrombocytopenia (platelet count <100,000/mm3), disorders of platelet function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Venous graft patency | At one year
  Venous graft patency as assessed by computed tomographic angiography or coronary angiography

SECONDARY OUTCOMES:
Major cardiac events (MACE) | At one year
  Acute myocardial infarction (AMI), Stroke, minor bleeding, death, rate of revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Hussein S Al-Amri, MD, Study Director — Prince Sultan Cardiac Center (PSCC), Riyadh
Locations (1):
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia